CLINICAL TRIAL: NCT05959551
Title: Modulating Functional Brain Connectivity Using High Definition Transcranial Direct Current Stimulation (HD-tDCS)
Brief Title: HD-tDCS to Modulate Connectivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HS24853
Record Dates: First submitted 2023-06-20; First posted 2023-07-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Electricity; Effects

STUDY DESIGN:
Intervention Model Description: 4 active treatment groups + 1 inactive treatment group
Who Masked: Participant
Masking Description: Randomization will happen after baseline assessment. After-intervention assessment will only consist of self-report and computerized assessment. Participants will not aware of the treatment group that they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- left DLPFC stimulation (Experimental): HD-tDCS will be used to deliver direct current to the target via rubber electrodes and HD-tDCS gels. The 9 electrodes (8 channels + 1 ground) positions and current intensity will be determined based on computer simulation using HDTargets software (Soterix Inc.) that results in maximum focal current on the left dorsolateral prefrontal cortex (DLPFC; x=-44, y=10, z=30) with inward field orientation. The peak current will not exceed 2 mA. A constant current will be delivered for 20 minutes.
  Interventions: Device: high definition transcranial direct current stimulation (HD-tDCS)
- right DLPFC stimulation (Experimental): HD-tDCS will be used to deliver direct current to the target via rubber electrodes and HD-tDCS gels. The 9 electrodes (8 channels + 1 ground) positions and current intensity will be determined based on computer simulation using HDTargets software (Soterix Inc.) that results in maximum focal current on the right dorsolateral prefrontal cortex (DLPFC; x=+42, y=+14, z=+30) with inward field orientation. The peak current will not exceed 2 mA. A constant current will be delivered for 20 minutes.
  Interventions: Device: high definition transcranial direct current stimulation (HD-tDCS)
- left IPL stimulation (Experimental): HD-tDCS will be used to deliver direct current to the target via rubber electrodes and HD-tDCS gels. The 9 electrodes (8 channels + 1 ground) positions and current intensity will be determined based on computer simulation using HDTargets software (Soterix Inc.) that results in maximum focal current on the left intraparietal lobe (IPL; x=-50, y=-36, z=+42) with inward field orientation. The peak current will not exceed 2 mA. A constant current will be delivered for 20 minutes.
  Interventions: Device: high definition transcranial direct current stimulation (HD-tDCS)
- VLPFC-PCC stimulation (Experimental): HD-tDCS will be used to deliver direct current to the target via rubber electrodes and HD-tDCS gels. The 9 electrodes (8 channels + 1 ground) positions and current intensity will be determined based on computer simulation using HDTargets software (Soterix Inc.) that results in maximum focal current on the left ventrolateral prefrontal cortex (VLPFC; x=-50, y=+26, z=+8) and posterior cingulate cortex (PCC; x=1, y=-61, z=38) with inward field orientation. The peak current will not exceed 2 mA. A constant current will be delivered for 20 minutes.
  Interventions: Device: high definition transcranial direct current stimulation (HD-tDCS)
- Sham stimulation (Sham Comparator): One of the above three targets will be randomly selected. The current will be applied for 30 seconds ramp-up followed by 30 seconds ramp-down.
  Interventions: Device: high definition transcranial direct current stimulation (HD-tDCS)

INTERVENTIONS:
Device: high definition transcranial direct current stimulation (HD-tDCS) — HD-tDCS will be provided for 20 minutes for each stimulation with peak intensity of 2mA.

SUMMARY:
The purpose of the proposed study is to broaden our understanding on the neural effects of High Definition Transcranial Direct Current Stimulation (HD-tDCS) so that its clinical effects can be further improved.

DETAILED DESCRIPTION:
Normal healthy individuals will be recruited and undergo a standardized neuropsychological assessment (ANAM, MoCA, BDI-II, ToMS, and MAAS) and magnetic resonance imaging (MRI). During MRI, HD-tDCS will be applied. Four different stimulation targets will be investigated, and subjects will be randomly assigned for each target groups or sham group. After HD-tDCS/MRI session, subjects will be re-assessed with standardized neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

- All other than excluded.

Exclusion Criteria:

* History or susceptibility to any neurological or psychiatric diseases, particularly seizures
* abnormal MRI
* metal implants or a cardiac pacemaker
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
change of functional connectivity | 0-11 minutes after the stimulation contrasting baseline (before stimulation)
  Changes in seed-based connectivity originating from the targeted brain regions immediately after the brain stimulation

SECONDARY OUTCOMES:
change of cerebral blood flow | 12-16 minutes after the stimulation contrasting baseline (before stimulation)
  Changes in Cerebral Blood Flow (estimated using pseudo continuous arterial spin labeling )
Toronto Mindfulness Scale (curiosity) | Baseline, then within 1-2 hours from stimulation
  mindfulness scale for curiosity. min: 0, max: 30. Higher score means higher curiosity-mindfulness.
Toronto Mindfulness Scale (decentering) | Baseline, then within 1-2 hours from stimulation
  mindfulness scale for decentering. min: 0, max: 35. Higher score means higher decentering-mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No